CLINICAL TRIAL: NCT03243643
Title: Tolerability, Safety, Pharmacokinetics and Efficacy of HS-10241 Single Agent or Combined With Apatinib in Patients With Advanced Solid Tumors
Acronym: HS:Hansoh;
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS-10241-I-101
Record Dates: First submitted 2017-07-18; First posted 2017-08-09 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-07

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-1024+apatinib (Experimental): For part 1 (PK study) subjects will be given single dose of HS-10241 and then multiple dose of HS-10241 (1 cycle, each cycle 14days) and then HS-10241+aptatinib (each cycle 21 days) until PD.
  For part 2 (expansion study) subjects will be given HS-10241+aptatinib (each cycle 21 days) until PD (Progression of disease).
  Interventions: Drug: HS-10241; Drug: Apatinib

INTERVENTIONS:
Drug: HS-10241 — HS-10241 is provided as white, film-coated,immediate release tablets containing HS-10241 at dosage strengths of 20mg/50mg/100 mg. Multiple tablets of HS-10241 will be administered daily to achieve targeted doses of HS-10241: 200 mg-1200 mg. Tablets will be orally administered with 240 ml water, once daily, 1 hour before/after a meal.
  Other Names: c-met inhibitor
Drug: Apatinib — Apatinib is provided as white, film-coated,immediate release tablets containing aptinib at dosage strengths of 250mg. Apatinib will be administered daily to achieve targeted doses of 500 mg. Tablets will be orally administered with 240 ml water, once daily, 1 hour before/after a meal.

SUMMARY:
To investigate tolerability, safety, pharmacokinetics and efficacy of C-met Kinase Inhibitor HS-10241 single agent or combined with Apatinib in Subjects With Advanced Solid Tumours that are not eligible for conventional or intensive treatment. The dose of HS-10241 will be escalated to determine the dose limiting toxicity (DLT) and the maximum tolerated dose (MTD) of HS-10241 single agent and in combination with Apatinib in advanced cancer patients. At the same time, pharmacokinetic characteristics and preliminary efficacy of HS-10241 or combined with Apatinb will be observed in advanced cancer patients. To determine the recommended dosage regimen for phase II.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age.
2. Histologically or cytologically confirmed advanced or metastatic solid tumor for which standard therapy does not exist, has failed.；For part 2 (Expansion part) c-met immunohistochemistry (IHC) positive（IHC++ or IHC+++）and with at least one measurable disease according to RECIST 1.1.
3. No difficulty that may hamper compliance and/or absorption of the tested product (swallowing difficulty, chronic gastrointestinal disease like diarrhea and intestinal obstruction )
4. ECOG (Eastern Cooperative Oncology Group) performance status of 0～1.
5. Life expectancy of at least 3 months.
6. Adequate organ function:（No blood transfusion or hematopoietic stimulating factor within 14days of screening stage）：
7. Acceptable hematologic status (without hematologic supports including hematopoietic factor, blood transfusion) defined below:：Absolute neutrophil count (ANC) ≥1500/μL
8. Platelet count ≥90000/μL,，Hemoglobin ≥9.0 g/dL
9. Acceptable liver function defined below:：Total bilirubin ≤ 1.5 times upper limit of normal range (ULN)
10. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times ULN; however, ≤5 times ULN in a subject who has liver metastases.
11. Acceptable renal function defined below:：Serum creatinine ≤1.5 times ULN or calculated creatinine clearance (by the Cockcroft-Gault formula) ≥60 mL/minutes.
12. Acceptable cardiac function defined below:： left ventricular ejection fraction，LVEF≥50% ；normal ECG，QTc male<450ms，female<470ms
13. Recovered from toxicities of prior anti-cancer treatment (NCI-CTCAE 4.03≤ grade 1, except alopecia); Proper period of wash out of previous treatment (at least 5 half-life wash out), e.g. No nitrosoureas or mitomycin within 6 weeks，no cytotoxic drugs, monoclonal antibodies, radiation therapy, or surgery within 4 weeks and no endocrine therapy or tyrosine kinase inhibitors (TKIs) within 2 weeks before first dose of the tested product.
14. Non-surgical sterilization or post-menopause female must agree to use effective means of contraception (IUD , medication or condom ) during and 8 weeks after the clinical trial.Human Chorionic Gonadotropin ( HCG ) serum test must be negative tested 7 days before the first dose of tested product and not being in the lactation period. For male subjects whose female partners have childbearing potential must be surgical sterilization or agree to use effective means of contraception during and 120 days after the clinical trial.
15. Tumor tissue sample available or agree to provide biopsies for testing.
16. Volunteer to participate in the clinical trial, understand the procedure of trial and approved informed consent obtained before entering the trial.

Exclusion Criteria:

1. Failed in previous c-met or VEGFR inhibitor treatment;
2. Participation in other clinical trial or the last dose of the other trail was taken within 4 weeks.
3. Other anti-cancer treatment might be received during the trial leading to pause of the trial.
4. Tumor infiltration of the vessel, tumor cavity or necrosis with risk of hemorrhage.
5. Central nervous system (CNS) metastases or meningeal metastases or primary nervous system tumor untreated by surgery or radiotherapy.
6. Patients with clinical symptoms of ascites or pleural effusion, need therapeutic puncture and drainage.
7. Uncontrolled chronic systematic complications (such as chronic pulmonary , hepatic, renal or cardiac diseases).
8. Grade II myocardial ischemia or myocardial infarction or uncontrolled arrhythmia. Cardiac dysfunction with New York Heart Association (NYHA) Class III or IV.
9. Hypertension and unable to be controlled within normal level following treatment of two anti-hypertension agents (systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥90 mmHg).
10. Urine protein≥ ++，or 24 hour urine protein≥1.0 g；
11. Patients with or previous with clinically significant hemorrhage within 3 months, with hemorrhage risk or being in anticoagulant and fibrinolytic treatment like gastrointestinal bleeding , hemorrhagic ulcers, baseline defecate occult blood positive and above or vasculitis. Abnormal coagulant function such as INR(international normalized ratio)>1.5 or PT （Prothrombin Time）>ULN+4 seconds）.
12. Arterial or venous thromboembolism events within 6 months，like cerebral vascular accident (transient ischemic attack, cerebral hemorrhage or cerebral infarction) or deep venous thrombosis and pulmonary embolism.
13. Active infection needed for treatment.
14. HIV,HBV (Hepatitis B Virus), HCV (Hepatitis C Virus) positive（HBV：HBsAg positive with hepatic function abnormality and HBV-DNA≧104 copy/mL，HCV：HCV-RNA positive with hepatic function abnormality）needed for antivirus treatment（only for Part 1）.
15. History of mental or neurological disorders.
16. Psychiatric drug abuse history or addiction history
17. Unable to complete the trial or withdraw in the middle of the trial due to conditions like psychological state, family relationship, social or geographical factors or with concomitant treatment or abnormal laboratory examinations judging by the investigator.
18. Concomitant diseases ( uncontrolled hypertension , severe diabetes and thyroid disease ) deemed by the investigator to be likely to interfere with the subjects safety or leads to discontinuation from the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Day1 to day 38 (DLT observation period)
  To assess MTD and DLT of HS-10241 single agent（D1-D17） then combined with aptatinib （D18-D38） in patients with advanced solid tumors.According to the "3+3" dose escalation design DLT will be determined.
Maximum Tolerated Dose (MTD) | Day1 to day 38 (DLT observation period)
  One dose level below the dose level determined as DLT will be MTD.

SECONDARY OUTCOMES:
Adverse events and Serious Adverse Events | From the day of ICF (Informed Consent Form) until 30 days after the last dose
  To asess the safety of HS-10241 single agent the combined with apatinib in patients with advanced solid tumor.
The measurement of maximum plasma concentration (Cmax) | Day 1 to day 38
  Including HS-10241 single dose （D1）/multiple dose of HS-10241（D17） and multiple dose of Apatinib（D38）.
The measurement of the area under the plasma concentration-time versus time curve(AUC) | Day 1 to day 38
  Area Under Curve(AUC0-t) will be measured after single dose administration of HS-10241 at day 1.AUC0-t and AUC0-inf are measured after repeated once-daily dose administration of HS-10241 at day 14.AUC0-t and AUC0-inf are measured after repeat once-daily dose administration of apatinib at day 38.
The measurement of the area under the plasma concentration-time versus time curve(AUC) | Day 1 to day 38
  AUC(0-inf) will be measured after single dose administration of HS-10241 at day 1.AUC0-t and AUC0-inf are measured after repeated once-daily dose administration of HS-10241 at day 14.AUC0-t and AUC0-inf are measured after repeat once-daily dose administration of apatinib at day 38.
The measurement of time of maximum plasma concentration (Tmax) | Day 1 to day 38
  Including HS-10241 single dose （D1）/multiple dose of HS-10241（D17） and multiple dose of apatinib（D38）.
The measurement of elimination half life (T1/2) | Day 1 to day 38
  T1/2 is measured after single dose administration of HS-10241 at day 1. T1/2 is measured after repeat once-daily dose administration of HS-10241 at day 17.
The Measurement of mean retention time (MRT) | Day 1 to day 38
  MRT is measured after single dose administration of HS-10241 at day 1.
The measurement of apparent volume of distribution (Vd) | Day 1 to day 38
  Vd is measured after single dose administration of HS-10241 at day 1. Vd is measured after repeated once-daily dose administration of HS-10241 at day 17.
The measurement of clearance (Cl) | Day 1 to day 38
  Vd is measured after single dose administration of HS-10241 at day 1. Vd is measured after repeated once-daily dose administration of HS-10241 at day 17.
Duration of Response Rate | Approximately 1 year
  Determined using RECIST v1.1 criteria
Progression-Free Survival | Approximately 1 year
  Determined using RECIST v1.1 criteria
Objective Response Rate | Approximately 1 year
  Determined using RECIST v1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chendu, China

IPD SHARING:
Plan to Share IPD: No